CLINICAL TRIAL: NCT00521261
Title: Immune Consolidation With Allogeneic Activated T Cells Armed With OKT3 x Rituxan (Anti-CD3 x Anti-CD20) Bispecific Antibody (CD20Bi) After Allogeneic Peripheral Blood Stem Cell Transplant for High Risk CD20+ Non-Hodgkin's Lymphoma (Phase I)
Brief Title: Donor T Cells, Low-Dose Aldesleukin, and Low-Dose GM-CSF After Donor Stem Cell Transplant in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000561787; P30CA022453 (NIH); WSU-2007-034; 2365-1186500223.02
Record Dates: First submitted 2007-08-24; First posted 2007-08-27 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Lymphoma
Keywords: recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult T-cell leukemia/lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; Waldenstrom macroglobulinemia; adult nasal type extranodal NK/T-cell lymphoma; recurrent adult grade III lymphomatoid granulomatosis; cutaneous B-cell non-Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, Extranodal NK-T-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: anti-CD3 x anti-CD20 bispecific antibody-armed activated T cells

SUMMARY:
RATIONALE: Giving high doses of chemotherapy before a donor stem cell transplant helps stop the growth of cancer cells. It also stops the patient's immune system from rejecting the donor's stem cells. Colony stimulating factors, such as aldesleukin and GM-CSF, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect). Giving an infusion of the donor's T cells that have been treated with antibodies after the transplant may help increase this effect. Sometimes the transplanted cells from a donor can also make an immune response against the body's normal cells. Giving tacrolimus and mycophenolate mofetil after transplant may stop this from happening.

PURPOSE: This phase I trial is studying the side effects and best dose of donor T cells given together with low-dose aldesleukin and low-dose GM-CSF after donor stem cell transplant in treating patients with relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of donor-derived allogeneic anti-CD3 X anti-CD20 bispecific antibody (CD20Bi)-armed activated T cells (ATC) when given with low-dose aldesleukin and low-dose sargramostim (GM-CSF) after allogeneic stem cell transplantation in patients with relapsed or refractory CD20-positive non-Hodgkin lymphoma.
* Perform trafficking studies using indium I 111-labeled unarmed ATC and ATC armed with CD20Bi in patients with evaluable lymphoma sites to determine whether armed ATC specifically traffic to tumor sites and correlate these data with CT and PET scans.
* Evaluate immune responses and immune reconstitution of T and B cells.

OUTLINE: All patients receive high-dose chemotherapy that is standard of care for their disease. Peripheral blood lymphocytes are obtained from the HLA-identical sibling donor and cultured to obtain activated T cells (ATC), some of which are subsequently armed with CD20 bispecific antibody (CD20Bi) and cryopreserved for later use. Patients then undergo allogeneic hematopoietic stem cell transplantation (SCT).

Patients receive ATC-CD20Bi IV on days 40, 70, 100, 130, and 160 after SCT. Patients receive low-dose aldesleukin subcutaneously (SC) once daily for 7 days beginning within 24 hours after each ATC-CD20Bi infusion and low-dose sargramostim (GM-CSF) SC every other day for 3 doses beginning within 24 hours after each infusion of ATC-CD20Bi. Patients also receive tacrolimus and mycophenolate mofetil as standard graft-vs-host disease prophylaxis. Treatment continues in the absence of unacceptable toxicity.

Some patients with well-defined or evaluable masses receive indium I 111 (^111I)-labeled ATC-CD20Bi IV and ^111I-labeled unarmed ATC and then undergo whole-body imaging for trafficking studies.

After completion of study treatment, patients are followed at 6 months, 12 months, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed CD20-positive non-Hodgkin lymphoma

  * Relapsed, resistant, or chemorefractory disease
* Must have an available HLA-identical sibling donor
* No significant skin breakdown from tumor or other disease

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* DLCO ≥ 50% of normal
* No symptomatic obstructive or restrictive pulmonary disease
* Creatinine ≤ 2.0 mg/dL OR creatinine clearance ≥ 60 mL/min
* Direct bilirubin ≤ 2.0 mg/dL (even if attributable to disease)
* SGOT and SGPT ≤ 2.5 times normal (even if attributable to disease)
* No history of severe hepatic dysfunction
* No severe cardiac dysfunction
* LVEF ≥ 50% by gated blood pool scan
* No major heart disease
* Patients with congenital or acquired heart disease or cardiac arrhythmias must undergo a cardiology consultation and evaluation
* No active infections

  * Patients who have not been seen and evaluated by a dentist for teeth cleaning and examination for potential sources of infection are ineligible
* HIV antibody negative
* No uncompensated major thyroid or adrenal dysfunction
* Not pregnant or nursing
* Persistently elevated systolic blood pressure (BP) ≥ 130 mm Hg or diastolic BP ≥ 80 mm Hg must be controlled with antihypertensive agents for at least 7 days prior to initiation of cell therapy

  * Patients with essential hypertension that is controlled with medication are eligible

PRIOR CONCURRENT THERAPY:

* Prior total dose of doxorubicin or daunorubicin must have been less than 450 mg/m^2 unless an endomyocardial biopsy shows less than grade 2 drug effect
* No concurrent nitroglycerin preparations for angina pectoris
* No antiarrhythmic drugs for major ventricular dysrhythmias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-10; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose
Time to relapse
Disease-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence G. Lum, MD, DSc, Principal Investigator — Barbara Ann Karmanos Cancer Institute